CLINICAL TRIAL: NCT05514002
Title: Randomized Participant- and Investigator-Blinded Trial to Compare the Clinical Efficacy of Recombinant Influenza Vaccine to Standard Dose Egg-Based Inactivated Influenza Vaccine Among Adults Aged 18-64 Years in the United States
Brief Title: Comparison of Recombinant Influenza Vaccine Versus Standard Egg-Based Inactivated Influenza Vaccine in Adults 18-64 Years
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funding.
Sponsor: Fatimah Dawood (U.S. Federal Agency)
Collaborators: Westat (Other); University of Arizona (Other); Florida A&M University (Other); Baylor College of Medicine (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Fatimah Dawood, Medical Officer, Principal Investigator, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0900f3eb81f9905e
Record Dates: First submitted 2022-08-08; First posted 2022-08-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Recombinant Influenza Vaccine (RIV) (Active Comparator)
  Interventions: Biological: Flublok Quadrivalent
- Standard-Dose Inactivate Influenza Vaccine (SD IIV) (Active Comparator)
  Interventions: Biological: Fluzone Quadrivalent

INTERVENTIONS:
Biological: Fluzone Quadrivalent — Intramuscular
  Arms: Standard-Dose Inactivate Influenza Vaccine (SD IIV)
Biological: Flublok Quadrivalent — Intramuscular
  Arms: Recombinant Influenza Vaccine (RIV)

SUMMARY:
This randomized, active comparator trial will compare the clinical efficacy of recombinant influenza vaccine (RIV) to standard-dose egg-based inactivated influenza vaccine (SD IIV) among adults aged 18-64 years. The primary study hypothesis is that the clinical efficacy of RIV is superior to that of SD IIV to prevent and attenuate influenza-like illness (ILI)-associated influenza virus infection. Relative efficacy will be assessed by comparing rates of ILI-associated reverse transcription polymerase chain reaction (RT-PCR)-confirmed influenza virus infection and measures of infection and illness attenuation among participants who receive RIV versus SD IIV. A secondary hypothesis is that humoral and cell-mediated immune responses to RIV are superior to responses to SD IIV. Relative immunogenicity will be assessed by comparing markers of humoral and cell-mediated immune responses post-vaccination among a subset of participants who receive RIV versus SD IIV.

DETAILED DESCRIPTION:
This randomized, active comparator trial will compare the clinical efficacy of recombinant influenza vaccine (RIV) to standard-dose egg-based inactivated influenza vaccine (SD IIV) among adults aged 18-64 years. The primary study hypothesis is that the clinical efficacy of RIV is superior to that of SD IIV to prevent and attenuate influenza-like illness (ILI)-associated influenza virus infection. Relative efficacy will be assessed by comparing rates of ILI-associated reverse transcription polymerase chain reaction (RT-PCR)-confirmed influenza virus infection and measures of infection and illness attenuation among participants who receive RIV versus SD IIV. A secondary hypothesis is that humoral and cell-mediated immune responses to RIV are superior to responses to SD IIV. Relative immunogenicity will be assessed by comparing markers of humoral and cell-mediated immune responses post-vaccination among a subset of participants who receive RIV versus SD IIV

The trial will be conducted at up to 6 sites in the United States during at least two influenza seasons (2022-23 and 2023-24). Stratified enrollment procedures will be used to enroll a representative mix of participants based on age (18-49 and 50-64 years). In addition, an enrollment quota will be used to enroll a minimum proportion of trial participants that self-identify as from a racial or ethnic group that has been historically underrepresented in clinical trials to optimize the racial and ethnic representativeness of the trial population compared to the US source population.

Eligible participants at each site will be randomized 1:1 to receive a single dose of RIV (Flublok® Quadrivalent by Sanofi Pasteur, 45µg of HA per strain) versus a single dose of SD IIV (Fluzone® Quadrivalent by Sanofi Pasteur, 15 µg of HA per strain) during approximately September through mid-November of 2022 or 2023. At a subset of sites, approximately 120 participants per trial season will be recruited and enrolled into an immunogenicity substudy with blood collection. All study vaccines are licensed for use in adults aged >18 years in the United States; RIV is licensed for adults aged >=18 years and SD IIV is licensed for persons aged >=6 months. Participants and study investigators will be blinded to study arm assignment. Designated study staff administering vaccines will be aware of study arm assignment and will not be involved with study surveillance to avoid involvement with measurement of study outcomes.

All participants will be followed with surveillance for ILI-associated RT-PCR-confirmed influenza virus infection. ILI will be defined as subjective (i.e., participant-reported) fever, cough, runny nose, or sore throat. Starting at enrollment, participants will respond to weekly text messages or emails asking about new onset of ILI symptoms to familiarize them with the electronic surveillance procedures and keep them engaged in the study prior to circulation of influenza viruses in the community. Once national and/or state influenza surveillance systems indicate that influenza viruses have begun circulating in the United States or no later than the first week of December, participants will also self-collect mid-turbinate nasal swabs (henceforth referred to as 'nasal swabs') with onset of ILI symptoms and self-ship or drop off swabs at designated sites for shipment to a central laboratory. Samples will be tested for influenza viruses by real-time reverse transcription polymerase chain reaction (RT-PCR). Samples may also be tested for Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) infection and other respiratory viruses. During the influenza virus circulation period or no later than the first week of December, participants who report ILI symptoms during the surveillance contacts will complete follow-up questionnaires to provide detailed information about their illnesses. Electronic surveillance and nasal swab collection will continue until local influenza virus circulation ends with the option to restart surveillance if additional periods of influenza virus circulation occur through May of each trial season.

Participants in the immunogenicity substudy will have blood collected just prior to vaccination and at approximately 7 days, 28 days, and 6 months post-vaccination to evaluate humoral and cell-mediated immune responses to vaccination; these participants will also have two nasal swabs collected prior to vaccination and at approximately 7 and 28 days post-vaccination for human microbiome characterization.

Sites will aim to enroll a combined total of up to 16,247 participants during the 2022-23 and 2023-24 seasons; up to about 7,000 of these will be in the first year. The immunogenicity substudy site(s) will aim to enroll 120 participants each season (60 per vaccine arm) who will contribute blood for serum, plasma, and peripheral blood mononuclear cell (PBMC) collection and nasal swabs for human microbiome characterization. A blinded sample size re-estimation will be conducted at the end of the first trial season by an independent designated statistician with experience with adaptive trial approaches. The analysis will follow a pre-specified analysis plan, and the recommended revised sample size will be shared with the trial steering committee for decision-making. Participants from the first trial season may be eligible for the second trial season; all participants will complete eligibility screening and consent processes at the start of each trial season. Participants from the first trial season who consent to participate in the second trial season will be rerandomized.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years
* Comfortable reading and responding to text messages or emails sent in either English, Spanish, or Chinese
* Currently enrolled as a student in a college or graduate degree program AND attending in-person classes with other students.

OR Currently employed as a frontline worker defined as an occupation that cannot be done from home or alone AND have direct face-to-face contact, defined as being within 6 feet, or about two arms' lengths, with co-workers, patients or the public as part of full-time (at least 20 hours per week) job responsibilities.

* Have daily access to the internet and a mobile phone that can send and receive text messages.
* Plan to continue to live/work in the study area through May 2023 (if trial season 1) or May 2024 (if trial season 2). For students in college or graduate degree programs, this is defined as living/working in the area excluding brief absences during school vacation periods.

Exclusion Criteria:

* Lives with another person who is already enrolled in this study as reported by the subject.
* Previous hypersensitivity reaction to the study vaccines as reported by the subject.
* Has already received current year influenza vaccine on our after July 1, 2022 as reported by the subject.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3988 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
ILI-associated RT-PCR-confirmed influenza virus infection | Through influenza season completion, approximately 16 weeks
  Time from 14 days post study influenza vaccination or the start of surveillance for influenza virus infection (whichever occurs later) to event

SECONDARY OUTCOMES:
ILI-associated RT-PCR-confirmed influenza virus infection by circulating virus subtypes and lineages | Through influenza season completion, approximately 16 weeks
  Time from 14 days post study influenza vaccination or the start of surveillance for influenza virus infection (whichever occurs later) to event
ILI-associated RT-PCR-confirmed influenza virus infection with vaccine and drifted strains (as feasible based on circulating viruses) | Through influenza season completion, approximately 16 weeks
  Time from 14 days post study influenza vaccination or the start of surveillance for influenza virus infection (whichever occurs later) to event
Time (in days) to return to usual health | Through ILI-associated RT-PCR-confirmed influenza virus infection episode completion, up to approximately 14 days
Mean highest overall symptom score and symptom score by days since symptom onset using the FLU-PRO© Plus questionnaire | Through ILI-associated RT-PCR-confirmed influenza virus infection episode completion, up to approximately 14 days
Duration (in days) of missed work or school influenza virus infections | Through ILI-associated RT-PCR-confirmed influenza virus infection episode completion, up to approximately 14 days
Geometric mean viral ribonucleic acid (RNA) load measured by quantitative PCR, as feasible | Through ILI-associated RT-PCR-confirmed influenza virus infection episode completion, up to approximately 14 days
HI (or MN as appropriate) responses to cell- and/or egg-grown vaccine reference viruses for each study season at approximately 28 days, and 6 months post-vaccination | At approximately 28 days and 6 months post-vaccination
  As measured by Geometric Mean Titer (GMT) ratio defined as the ratio of GMTs between study arms and Seroconversion rate (SCR) defined as the proportion of participants with paired samples that achieved ≥ 4 fold rises comparing post- versus pre-vaccination titers, and achieving post vaccination titers ≥ 40

OTHER OUTCOMES:
GMT by NAI and antibody dependent cellular cytotoxicity function assays pre- and post- vaccination | At approximately 28 days and 6 months post-vaccination
Percentage and absolute number of class switched B cells that are plasmablasts (CD38hi, CD27hi, CD71hi) | At approximately 7 and 28 days and 6 months post-vaccination
Percentage of vaccine HA specific antibody secreting cells pre- and post-vaccination | At approximately 7 and 28 days and 6 months post-vaccination
Percentage and absolute numbers of selected immunologic measures as described below | At approximately 7 and 28 days and 6 months post-vaccination
  Immunologic measures including IgG and IgA B cells that bind the vaccine HA, CD4+ and CD8+ T cells per ml of selected phenotypes, and influenza-specific CD8+ T cells degranulating during stimulation (CD107A) and producing IFN-γ, TNF-α, IL-2, and/or granzyme B as measured by intracellular cytokine staining pre- and post-vaccination
Number and frequencies of influenza-specific CD4+ T cells producing IFN-γ (Th1), IL-4 (Th2), IL-17 (Th17), and CD40L (after subtracting background levels of cytokine production/activation marker expression) by intracellular cytokine staining. | At approximately 7 and 28 days and 6 months post-vaccination
Number of OX40+ CD25+ activated CD4+ or CD8+ T cells post-vaccination (after subtracting background levels of cytokine production/activation marker expression) by activation induced marker assays. | At approximately 7 and 28 days and 6 months post-vaccination
B and T cell repertoires in a subset of subjects | At approximately 7 and 28 days and 6 months post-vaccination
Frequencies of natural killer cells and innate lymphoid cell subsets | At approximately 7 and 28 days and 6 months post-vaccination
RT-PCR-confirmed SARS-CoV-2 infections per 10,000 person-weeks | Through SARS-CoV-2 virus circulation period completion, up to approximately 16 weeks
Reverse-transcription polymerase chain reaction (RT-PCR)-confirmed SARS-CoV-2 infection (as feasible during trial seasons when SARS-CoV-2 testing is done) | Through SARS-CoV-2 virus circulation period completion, up to approximately 16 weeks
  Time from 7 days post booster COVID-19 vaccination or 14 days post primary series COVID-19 vaccination to event

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah S Dawood, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - Florida A&M University, Tallahassee, Florida
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Upon the completion of all study deliverables and after a suitable moratorium, external parties may request de-identified study data from the steering committee as specified in U.S. Government Data Sharing guidelines.
Supporting Information: Study Protocol
Time Frame: Upon the completion of all study deliverables and dissemination of analyses to meet the protocol objectives.

REFERENCES:
- [Derived] Grant L, Whitaker JA, Yoon SK, Lutrick K, Bhargava S, Brown CP, Zaragoza E, Fink RV, Meece J, Wielgosz K, El Sahly H, Hegmann KT, Lowe AA, Southworth A, Tatum T, Ball SW, Levine MZ, Thiese MS, Battan-Wraith S, Barnes J, Phillips AL, Fry AM, Dawood FS; Randomized Assessment of Influenza Vaccine Efficacy Network (RAIVEN). Relative Effectiveness and Immunogenicity of Quadrivalent Recombinant Influenza Vaccine Versus Egg-Based Inactivated Influenza Vaccine Among Adults Aged 18-64 Years: Results and Experience From a Randomized, Double-Blind Trial. Open Forum Infect Dis. 2024 Sep 26;11(10):ofae559. doi: 10.1093/ofid/ofae559. eCollection 2024 Oct. PMID 39416990